CLINICAL TRIAL: NCT04825431
Title: A Phase 1 Open-label Study Evaluating the Pharmacokinetics and Mass Balance of [14C] TAS-205 in Healthy Volunteers
Brief Title: Mass Balance Study of [14C] TAS-205 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10053070
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — TAS-205

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-205, [14C]TAS-205 (Experimental)
  Interventions: Drug: TAS-205, [14C]TAS-205

INTERVENTIONS:
Drug: TAS-205, [14C]TAS-205 — single oral administration under fasted conditions on day 1

SUMMARY:
To evaluate the pharmacokinetics, mass balance recovery, metabolite profile and metabolite identification of [14C]TAS-205 following oral single doses.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy adult male who provided written informed consent to participate in the study
2. Aged 20 years or older and younger than 40 years at the time of informed consent
3. Capable of oral intake.
4. Body weight of 50 kg or more and body mass index of 18.5 or more and less than 25.0

Key Exclusion Criteria

1. Had current or previous hypersensitivity or allergy to drugs
2. Had current or previous drug abuse (including use of illicit drugs) or alcoholism
3. Had any concurrent disease (including symptoms and signs; however, diseases that do not affect valuations in the study such as asymptomatic pollinosis and wart are excluded)
4. Consumed foods or beverages containing the St. John's Wort within 28 days before study drug administration
5. Had blood pressure, pulse rate, and body temperature meeting any of the following at screening:

Systolic blood pressure: <90 mmHg or ≥140 mmHg, Diastolic blood pressure: <40 mmHg or ≥90 mmHg, Pulse rate: <40 beats per minute (bpm) or ≥100 bp, Body temperature: 35.0°C or ≥37.1°C

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2022-05-27 (Actual)

PRIMARY OUTCOMES:
Concentrations of total radioactivity in blood and plasma, plasma TAS-205 concentrations and the pharmacokinetics parameters of TAS-205 | Day 1 to Day 8
Radioactivity excretion and excretion rate，cumulative excretion, cumulative excretion rate into urine and feces. | Day 1 to Day 8
Radioactivity excretion and excretion rate，cumulative excretion, cumulative excretion rate in all excreta (urine and feces). | Day 1 to Day 8
Plasma, urinary, and fecal metabolite profiles of TAS-205 , and structural estimation. | Day 1 to Day 8

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Data will not be shared according to the Sponsor policy on data sharing. Taiho policy on data sharing may be found at https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html.

REFERENCES:
- [Derived] Hanada R, Takenaka T. Phase 1 Mass Balance Study of Pizuglanstat: An Investigational Hematopoietic Prostaglandin D Synthase Inhibitor. Clin Pharmacol Drug Dev. 2025 Mar;14(3):200-208. doi: 10.1002/cpdd.1504. Epub 2025 Jan 22. PMID 39840517